CLINICAL TRIAL: NCT06212544
Title: Strengthening Community Responses to Economic Vulnerability and HIV Inequities
Brief Title: An HIV Status-neutral Microeconomic Intervention
Acronym: Secure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Kristi Gamarel, Associate Professor of Health Behavior and Health Education, University of Michigan
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: F00423; R34MH130207 (NIH)
Record Dates: First submitted 2023-12-20; First posted 2024-01-19 (Actual); Results first posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Feasibility Studies
Keywords: Transgender; HIV; microeconomic

STUDY DESIGN:
Intervention Model Description: Pilot waitlist randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Intervention (Experimental): The intervention condition builds on our community partners' existing microeconomic intervention of: (1) a one-time emergency cash grant and (2) peer and legal support to obtain legal gender affirmation - plus a 12-week microeconomic intervention that adds: (3) weekly educational sessions and HIV prevention; (4) community mentoring; and (5) weekly posts of job openings in Detroit; and (6) a micro-grant for use towards acquiring self-led or formal employment
  Interventions: Behavioral: Immediate Intervention
- Delayed Arm (Active Comparator): Participants randomized to the control condition will receive UC during the 12-week period following randomization. Usual care consists of emergency assistance and access to legal name/gender marker change. After the RCT follow-up period is complete, waitlist control participants will be offered delayed access to the same intervention that is provided immediately to intervention arm participants.
  Interventions: Behavioral: Delayed Intervention

INTERVENTIONS:
Behavioral: Immediate Intervention — Enhanced microeconomic intervention
  Arms: Immediate Intervention
Behavioral: Delayed Intervention — Usual care and then access to enhanced microeconomic intervention
  Arms: Delayed Arm

SUMMARY:
The aim is the current study is to establish feasibility and acceptability of the SeCuRE intervention to improve HIV prevention and care continua outcomes. To meet this aim, the study has the following objectives:

1. To deliver a two-armed pilot RCT of the SeCuRE intervention with 40 transgender women of color.
2. The determine acceptability of the intervention with transgender women of color.

DETAILED DESCRIPTION:
This is a two-arm randomized waitlist controlled trial in which transgender women of color will be randomly allocated to either the enhanced microeconomic intervention that builds on the Trans Sistas of Color Project's existing microeconomic interventions, which includes: (1) $250 in emergency assistance; and (2) peer support to obtain legal gender affirmation (i.e., legal name and gender markers on identification documents). The existing intervention will be enhanced to include (1) 12 weekly educational group sessions on economic empowerment (i.e., job acquisition, income generation through micro-business, and financial literacy) and HIV prevention and care; (2) employment-focused mentoring; and (3) an unconditional grant ($1,200) for use towards acquiring self-led or formal employment. Each condition will complete a baseline survey prior to randomization, a follow-up survey immediately following intervention completion, and 3-month survey after intervention completion. Participants will also complete qualitative exit interviews within one month of completion of intervention completion for both conditions.

ELIGIBILITY:
Inclusion Criteria:

1. at least 18 years old;
2. assigned male at birth;
3. self identifies as female, transgender woman, or another feminine gender identity;
4. self identifies as a person of color (i.e., any racial/ethnic identity except non-Hispanic white);
5. reports earning less than $32,800 gross annual income (current living wage in Michigan);
6. reports condomless sex in the past 6 months;
7. lives in Detroit, MI greater metropolitan area (~50 mile radius);
8. speaks English.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2024-06-07 (Actual); Primary Completion 2025-02-26 (Actual); Study Completion 2025-02-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristi Gamarel, PhD, Principal Investigator — University of Michigan
Locations (1):
- Ruth Ellis Center, Highland Park, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
The investigators plan to share de-identified data per guidelines; however, data will be in aggregate form to ensure individuals are not identified in anyway.

REFERENCES:
- [Derived] Gamarel K, Mayo-Wilson LJ, Jadwin-Cakmak L, Reyes L, Monro D, Ubong IA, Sullivan S, Abad J, Poindexter J, Harris H, Riser C, Stephenson J, Ortiz G, Peitzmeier SM, Neilands TB, Poteat T. Strengthening Community Responses to Economic vulnerability (SeCuRE): a protocol of an HIV status-neutral pilot randomized clinical trial with transgender women of color in Detroit, Michigan. Pilot Feasibility Stud. 2024 Nov 8;10(1):135. doi: 10.1186/s40814-024-01558-5. PMID 39511631

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Immediate Intervention | Delayed Arm
Started | 19 | 20
Completed | 19 | 15
Not Completed | 0 | 5

BASELINE CHARACTERISTICS:
Population: The analytic sample is the same as the enrolled participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Immediate Intervention | Delayed Arm | Total
Number analyzed (Participants) | 19 | 20 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.2 (9.2) | 32.5 (6.6) | 32.8 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 20 | 39
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 16 | 18 | 34
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 18 | 33
  White | 0 | 0 | 0
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 19 | 20 | 39

OUTCOME MEASURES:

1. Primary Outcome: Acceptability Quantitative
Description: The Client Satisfaction Questionnaire (CSQ-8) will be used to assess intervention satisfaction. This is an 8-item scale where each individual item is scored separately with a range of 1 to 4 and a score of 3 or 4 on each item will be considered indicative of acceptable.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Intervention | Delayed Arm
Number analyzed (Participants) | 19 | 20
score on a scale | 3.9 (0.3) | 3.8 (0.7)
Statistical Analysis 1: Comparison: Immediate Intervention; Test type: Superiority; p < 0.05, ANOVA

ADVERSE EVENTS:
Time Frame: 6 month time period
Description: There were no adverse events reported.
Arm/Group | Immediate Intervention | Delayed Arm
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/20
Other Adverse Events (participants affected / at risk) | 0/19 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-04-10): https://cdn.clinicaltrials.gov/large-docs/44/NCT06212544/Prot_SAP_000.pdf
  • Informed Consent Form (2023-08-03): https://cdn.clinicaltrials.gov/large-docs/44/NCT06212544/ICF_001.pdf